CLINICAL TRIAL: NCT00490984
Title: Tongue Advancement for Obstructive Sleep Apnea. An Evaluation fo the Aspire Medical Advance System.
Brief Title: Tongue Advancement for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspire Medical (Industry)
Responsible Party: Jafar Shenasa, Director, Clinical and Regulatory Affairs, Aspire Medical, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS 001
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: obstructive sleep apena; tongue; surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Aspire Medical Advance System — The treatment includes a device that is surgically implanted in the tongue and lower jaw. The purpose of the implant is to prevent obstruction of the upper airway thereby improving breathing during sleep.

SUMMARY:
The objective of this study is to assess the feasibility, safety and effectiveness of tongue stabilization using Aspire Medical Advance™ System for the treatment of obstructive sleep apnea (OSA). Success is defined as a statistically significant reduction in AHI measured by polysomnography (PSG) from baseline to 6 months.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a major health problem in the United States and can result in excessive daytime sleepiness and cardiovascular problems. The primary treatment for OSA today is continuous positive airway pressure (CPAP). Many patients however are unable to tolerate sleeping with a CPAP machine. Surgery is one of the main treatment options available today to these CPAP-intolerant patients. However, current methods of sleep surgery are painful, morbid, and/or lack decent effectiveness.

This trial will measure the effectiveness of the Advance System, an implantable medical device to treat OSA. In the trial, patients who meet the study entry criteria receive a baseline sleep study (PSG). The Advance System is then implanted and 6 months after implantation, another PSG is performed. The trial will compare the baseline and the 6 month apnea-hypopnea indices

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of obstructive sleep apnea with AHI 15-50 measured within a year prior to enrollment with no major change in BMI
* Bewteen 20 and 65 years old
* Body Mass Index (BMI) ≤ 32
* Patient has been offered CPAP and has refused or failed to continue CPAP treatment
* Identified evidence of airway collapse, primarily at the base of the tongue
* Signed informed consent to participate in this clinical study

Exclusion Criteria:

* Prior OSA surgery except tonsillectomy, nasal surgery and uvulopalatopharyngoplasty; no airway surgery within 3 months prior to enrollment.
* Airway collapse at the level of the soft palate (palatal collapse).
* Enlarged tonsils (3+ and 4+)
* Anatomy unable to accommodate the implant
* Severe mandibular deficiency/retrognathia
* Unable and/or not willing to comply with treatment follow-up requirements.
* Pregnancy. (Female subjects of childbearing potential must have a negative pregnancy test prior to enrollment and should maintain adequate contraception during the study)
* Breastfeeding women
* Active systemic infection
* Allergy to any medication used during implantation
* Previous history of neck or upper respiratory tract cancer
* History of radiation therapy to neck or upper respiratory tract
* Dysphagia
* Major cardiovascular and pulmonary disorders
* Other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment and the procedures and evaluations pre- and post-treatment
* Enrollment in another pharmacological or medical device study that may effect or bias the results of this clinical study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Demonstrate the feasibility of tongue stabilization using the Advance™ System. Product implantation and stabilization of the tongue using the Advance™system will be measured by Pharyngoscopy and Cephalogram | 3 months
Evaluate the safety of the Advance™ System 3 Months after implantation. | 3 months
Compare baseline and 6 month apnea-hypopnea indices as measured by PSG studies. | 6 months

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) measured at 3 Months post-implantation | 3 months
Functional Outcomes of Sleep Questionnaire (FOSQ) measured at 3 Months post-implantation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris A. Stuck, MD, Principal Investigator — Deparment of Otorhinolaryngology, Head and Neck Surgery, University Hospital Mannheim; Evert Hamans, MD, Principal Investigator — Department of Otorhinolaryngology, University Hospital Antwerp
Locations (3):
- Universitair Ziekenhuis Antwerpen, Egedem, Belgium
- LENTE, Pilsen, Czechia
- University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- See also: Sponsor's web site; has basic product & patient information — http://www.aspiremedical.com/clinic_ous.html